CLINICAL TRIAL: NCT01665196
Title: Evaluation of 18F-FDG PET/CT in Diagnosis and Response Assessment of Patients With IgG4-Related Disease
Brief Title: 18F-FDG PET/CT for IgG4-Related Disease
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Zhaohui Zhu, Professor, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IgG4RD-PET
Record Dates: First submitted 2012-08-13; First posted 2012-08-15 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Autoimmune Disease
Keywords: IgG4-related disease; IgG4-RD; 18F-FDG; PET/CT
MeSH Terms: conditions — Autoimmune Diseases; Immunoglobulin G4-Related Disease | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 18F-FDG PET/CT scanning (Experimental): 18F-FDG PET/CT scanning will be performed in patients with IgG4RD to determine the pictorial characteristics and measure the standardized uptake values (SUVs) of the lesions and their response to treatment.
  Interventions: Drug: 18F-FDG

INTERVENTIONS:
Drug: 18F-FDG — Intravenous injection of single dose of 18F-FDG before treatment and after 4-week treatment, respectively.
  Other Names: 18F-Fluorodeoxyglucose; 2-Fluoro-2-deoxy-D-glucose; Fluorine-18-fluorodeoxyglucose

SUMMARY:
This is an open-label study to investigate the diagnostic performance of 18F-FDG PET/CT (positron emission tomography/computed tomography) in evaluation of patients with IgG4-related disease. A single dose of 18F-FDG will be intravenously injected into patients with IgG4-related disease before and after treatment.

DETAILED DESCRIPTION:
Immunoglobulin G4-related disease (IgG4-RD) is a recently defined emerging clinical entity characterized by tissue infiltration by IgG4-positive plasma cells, tissue fibrosclerosis and elevated serum IgG4 concentration. The most important feature of IgG4-RD is chronic inflammation with multiple organ involvement. However, some organ involvements are difficult to find by ultrasound, CT or MRI.

18F-FDG PET/CT is a sensitive imaging tool for inflammation. In this study, PET/CT were performed in patients with IgG4-RD both before and after glucocorticoid treatment by a single dose of 18F-FDG. Visual and semiquantitative method will be employed to assess the PET/CT images. The PET/CT image data will be used to establish a diagnostic model as well as assessment criteria for response evaluation of IgG4-RD treatments.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Age 18-75 years old with informed consent
* Patients with IgG4-RD:

  1. swelling, sclerosing and inflammatory involvement of one or more organ, including sclerosing pancreatitis, sclerosing cholangitis, inflammatory pseudotumors, retroperitoneal or mediastinal fibrosis, interstitial nephritis, hypophysitis, sclerosing dacryoadenitis, sialadenitis, inflammatory aortic aneurysm, lymphadenopathy, or other inflammatory conditions;
  2. elevated serum IgG4 (>1.35 g/L) or with histopathologic features of fibrosis and/or lymphocytic and polyclonal plasma cell infiltration (and IgG4+ plasma cells on immunohistology when performed);
  3. exclusion of other diseases.

Exclusion Criteria:

* Females planning to bear a child recently or with childbearing potential;
* Inability to complete the examination;
* Concurrent severe and/or uncontrolled and/or unstable diseases;
* Currently under treatment using glucocorticoids.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-09; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Visual analysis of organ involvement and treatment response of the IgG4-RD patients. | 1 year
  Visual analysis will be performed by consensus reading by at least 3 experienced nuclear medicine physician. The 18F-FDG PET/CT pattern of IgG4-RG will be extracted and summarized. The response to anti-immune treatment will be assessed.

SECONDARY OUTCOMES:
Semiquantitative measurement of lesion metabolism and treatment response of the IgG4-RD patients. | 1 year
  The semiquantitative analysis will be performed by measuring the standardized uptake values (SUVs) of 18F-FDG by the IgG4-RD lesions and calculate the SUV changes before and after anti-immune treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Wen Zhang, MD, Study Director — Deptment of Rheumatology, Peking Union Medical College Hospital; Fang Li, MD, Study Chair — Department of Nuclear Medicine, Peking Union Medical College Hospital, CAMS & PUMC; Zhaohui Zhu, MD, Principal Investigator — Department of Nuclear Medicine, Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang J, Chen H, Ma Y, Xiao Y, Niu N, Lin W, Wang X, Liang Z, Zhang F, Li F, Zhang W, Zhu Z. Characterizing IgG4-related disease with (1)(8)F-FDG PET/CT: a prospective cohort study. Eur J Nucl Med Mol Imaging. 2014 Aug;41(8):1624-34. doi: 10.1007/s00259-014-2729-3. Epub 2014 Apr 25. PMID 24764034